CLINICAL TRIAL: NCT01352507
Title: An Evaluation of Tadalafil and Sildenafil Treatment in Men With Erectile Dysfunction in China
Brief Title: A Study of Tadalafil and Sildenafil in Men With Erectile Dysfunction in China
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 14035; H6D-CR-LVIZ (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-05-10; First posted 2011-05-12 (Estimated); Results first posted 2013-04-26 (Estimated); Last update posted 2013-04-26 (Estimated); Status verified 2013-03

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — Tadalafil; Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tadalafil then Sildenafil (Experimental): 20 mg tadalafil taken orally, as needed, for 8 weeks, followed by 100 mg sildenafil taken orally, as needed, for an additional 8 weeks. There is a washout period of 7-10 days between treatments.
  At the end of the two 8-week treatment periods, participants will be allowed to enter an 8-week extension phase on their preferred medication for erectile dysfunction (ED).
  Interventions: Drug: Tadalafil; Drug: Sildenafil
- Sildenafil then Tadalafil (Active Comparator): 100 mg sildenafil taken orally, as needed, for 8 weeks, followed by 20 mg tadalafil taken orally, as needed, for an additional 8 weeks. There is a washout period of 7-10 days between treatments.
  At the end of the two 8-week treatment periods, participants will be allowed to enter an 8-week extension phase on their preferred medication for ED.
  Interventions: Drug: Tadalafil; Drug: Sildenafil

INTERVENTIONS:
Drug: Tadalafil — Administered Orally
  Other Names: Cialis; LY450190
Drug: Sildenafil — Administered Orally

SUMMARY:
The primary objective of this study is to evaluate whether, after two 8-week treatment periods, male patients with erectile dysfunction (ED) in China prefer 20 milligram (mg) tadalafil or 100 mg sildenafil. This trial consists of two treatment periods of 8 weeks each and an extension phase of 8 weeks, for a total of 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

Study Subjects

* Are able to read, understand and provide signed informed consent.
* Have a history ED of any etiological classification (psychogenic, organic, or mixed) and any severity for at least 3 months.
* Have never taken any phosphodiesterase 5 (PDE5) inhibitor for the treatment of ED.
* Anticipate having the same female sexual partner during the study for recording responses to efficacy questionnaires. If a qualifying participant has more than one female partner during the study, the participant will not be excluded from the trial. However, the participant will be required to respond to the questionnaires based on his sexual interactions with only one of these partners.
* Make at least 4 sexual intercourse attempts, with the female sexual study partner, during the 4-week run-in period and during the final 4 weeks of each 8-week treatment period.
* Not use any ED treatment including the use of herbal therapy and traditional Chinese medicine (TCM) for the treatment of ED other than study medication at any time during the study and for 96 hours after study completion.

Partners

* Are female, at least 18 years of age at screening and will have the same male study subject as her sexual partner during the study.
* Are able to read, understand and provide signed informed consent.
* Agree to make at least 4 sexual intercourse attempts with the male sexual study partner during the 4-week run-in phase and during the final 4 weeks of each 8-week treatment period.
* Willing to participate in recording responses to efficacy questionnaires, sexual quality of life questionnaires and other instruments used in this study.

Exclusion Criteria:

* Present with ED caused by other primary sexual disorders including premature ejaculation or ED caused by untreated endocrine disease.
* Have a history of radical prostatectomy, or other pelvic surgery with subsequent failure to achieve erection.
* Have a history of penile implant.
* Have a clinically significant penile deformity in the opinion of the investigator.
* Exhibit evidence of clinically significant renal insufficiency as determined by the investigator, or defined as receiving renal dialysis or having an estimated creatinine clearance of less than (<)30 milliliters per minute (mL/minute) at screening, as calculated by the local laboratory using the Cockcroft-Gault formula.
* Exhibit evidence of active symptomatic hepatobiliary disease at Visit 1.
* Exhibit Hemoglobin A1c greater than (>) 11 percent (%) at screening, in patients with a history of diabetes mellitus of any type.
* Present with chronic stable angina treated with long-acting nitrates, or with chronic stable angina requiring short-acting nitrates in the last 90 days, or with angina occurring during sexual intercourse in the last 6 months.
* Have met the criteria for unstable angina within 6 months before screening, or have a history of myocardial infarction or coronary artery bypass graft surgery within 90 days before screening, or percutaneous coronary intervention within 90 days before screening.
* Have any supraventricular arrhythmia with an uncontrolled ventricular response (mean heart rate >100 bpm) at rest, or have any history of spontaneous or induced sustained ventricular tachycardia (heart rate >100 beats per minute (bpm) for greater than or equal [≥] to 30 seconds) despite medical or device therapy, or use an internal cardioverter-defibrillator.
* Have a history of sudden cardiac arrest despite medical or device therapy.
* Exhibit any evidence of congestive heart failure within 6 months before screening.
* Have had a new or significant cardiac conduction defect within 90 days before screening.
* Exhibit systolic blood pressure >170 or <90 milliliters of mercury (mm Hg) or diastolic blood pressure >100 or <50 mm Hg at screening, or have a history of malignant hypertension.
* Have retinitis pigmentosa.
* Have a history of significant central nervous system injuries (including stroke and spinal cord injury) within the last 6 months.
* Have a history of human immunodeficiency virus (HIV) infection.
* Have a condition that in the opinion of the investigator would interfere with the patient's ability to provide informed consent or comply with study instructions, would place the patient at increased risk, or might confound the interpretation of study results.
* Currently receive treatment with nitrates, alpha [1]-adrenergic blockers (such as doxazosin), cancer chemotherapy, or antiandrogens (except finasteride taken as Propecia™ or Proscar® or Avodart® [dutasteride]).
* Have a history of drug, alcohol, or substance abuse within the past 6 months, as assessed by the investigator.
* Have received treatment within the last 30 days with a drug that has not received regulatory approval for any indication at the time of study entry.
* Patients who are currently taking TCM for ED treatment within the last 30 days prior to study entry or planned concomitant administration of TCM for ED treatment during study enrolment.
* Are currently enrolled in, or discontinued with the last 30 days from a clinical trial involving an investigational product or unapproved use of a drug or device, or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study. Patients who have been screen failures in other studies may be eligible if they satisfy the inclusion/exclusion criteria.
* Have a history of loss of vision in one eye because of non-arteritic anterior ischemic optic neuropathy (NAION), regardless of whether this episode was in connection or not with previous PDE5 inhibitor exposure.
* Have rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption lactose intolerance.
* Are currently in a sexual relationship with a female of child-bearing potential where no form of birth control is being used. A female of child-bearing potential is a female who is not surgically or chemically sterilized and who is between menarche and 1-year post menopause.
* Are currently in or are planning to be in a sexual relationship with a pregnant female or are currently in a relationship where either partner is actively trying to conceive.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 383 (Actual)
Dates: Start 2011-06; Primary Completion 2012-06 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (9):
- China (9):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beijing
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Changsha
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hangzhou
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nanjing
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shanghai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shenzhen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tianjin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wuhan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Xi'an

RESULTS

PARTICIPANT FLOW:
Groups:
- Tadalafil Then Sildenafil: 20 milligrams (mg) tadalafil taken orally, as needed, for 8 weeks, followed by 100 mg sildenafil taken orally, as needed, for an additional 8 weeks. There was a washout period of 7 to 10 days between treatments.
  At the end of the two 8-week treatment periods, participants were allowed to enter an 8-week extension phase on their preferred medication for erectile dysfunction (ED).
- Sildenafil Then Tadalafil: 100 mg sildenafil taken orally, as needed, for 8 weeks, followed by 20 mg tadalafil taken orally, as needed, for an additional 8 weeks. There was a washout period of 7 to 10 days between treatments.
  At the end of the two 8-week treatment periods, participants were allowed to enter an 8-week extension phase on their preferred medication for ED.
Period: Treatment Period 1
Arm/Group | Tadalafil Then Sildenafil | Sildenafil Then Tadalafil
Started | 190 | 193
Received Treatment | 182 | 188
Completed | 176 | 184
Not Completed | 14 | 9
Not completed — Adverse Event | 3 | 0
Not completed — Lost to Follow-up | 3 | 4
Not completed — Withdrawal by Subject | 7 | 5
Not completed — Physician Decision | 1 | 0
Period: Washout Period
Arm/Group | Tadalafil Then Sildenafil | Sildenafil Then Tadalafil
Started | 176 | 184
Completed | 176 | 183
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Treatment Period 2
Arm/Group | Tadalafil Then Sildenafil | Sildenafil Then Tadalafil
Started | 176 | 183
Received Treatment | 173 | 181
Completed | 170 (Six participants who completed Treatment Period 2 chose not to enter the Extension Phase.) | 180 (Seven participants who completed Treatment Period 2 chose not to enter the Extension Phase.)
Not Completed | 6 | 3
Not completed — Entry Criteria Not Met | 1 | 0
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Lack of Efficacy | 1 | 0
Period: Extension Phase
Arm/Group | Tadalafil Then Sildenafil | Sildenafil Then Tadalafil
Started | 164 | 173
Completed | 164 | 173
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tadalafil Then Sildenafil | Sildenafil Then Tadalafil | Total
Number analyzed (Participants) | 190 | 193 | 383
Age Continuous [Mean (Standard Deviation); unit: years] | 39.20 (10.52) | 40.66 (11.44) | 39.94 (11.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 190 | 193 | 383
Race/Ethnicity, Customized [Number; unit: participants]
  Chinese | 190 | 193 | 383
Region of Enrollment [Number; unit: participants]
  China | 190 | 193 | 383
International Index of Erectile Function (IIEF) Erectile Function (EF) Domain [Mean (Standard Deviation); unit: units on a scale] — IIEF-EF was the sum of Questions (Q)1 through 5 and Q15 of the IIEF. Q1 to Q5 were scored 0 (low/no erectile function) to 5 (high erectile function) and Q15 was scored 1 (no/low confidence) to 5 (high confidence). IIEF-EF domain scores ranged from 1 to 30. Higher scores represented better erectile function.
  units on a scale | 13.77 (5.37) | 14.19 (6.08) | 13.98 (5.73)
Erectile Dysfunction (ED) Severity [Number; unit: participants] — Investigator-reported severity of a participant's ED. ED was defined as a consistent change in the quality of erection adversely affecting participant satisfaction with sexual intercourse. Severity was based on investigator opinion.
  participants
    Mild | 63 | 68 | 131
    Moderate | 68 | 65 | 133
    Severe | 59 | 60 | 119
ED Duration [Number; unit: participants]
  ≥3 months to <1 year | 77 | 87 | 164
  ≥1 year | 113 | 106 | 219
ED Etiology [Number; unit: participants]
  Psychogenic | 46 | 41 | 87
  Organic | 11 | 13 | 24
  Mixed | 133 | 139 | 272

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Preferring Tadalafil Over Sildenafil Measured at Week 18 Using Question 1 of the "Phosphodiesterase 5 Inhibitor Treatment Preference" Questionnaire (PITPQ)
Description: PITPQ Question (Q) 1 was a dichotomous outcome measure in which the participant selected his preferred study treatment (tadalafil or sildenafil) to receive during the Extension Phase.
Time Frame: Week 18
Population: Randomized participants who completed both treatment periods (Week 18), responded to the PITPQ, and were analyzed according to their assigned treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- All Randomized Participants: Includes participants randomized to initially receive tadalafil (20 mg taken orally, as needed, for 8 weeks) and participants randomized to initially receive sildenafil (100 mg taken orally, as needed, for 8 weeks).
Arm/Group | All Randomized Participants
Number analyzed (Participants) | 350
percentage of participants | 69.1 [64 to 74]
Statistical Analysis 1: Comparison: All Randomized Participants; Null hypothesis (H0): The proportion of participants who chose tadalafil over sildenafil is equal to 0.5 (p = 0.5), versus alternative hypothesis (H1): p is not equal to 0.5 (2-sided test); Test type: Superiority or Other; p < 0.001, Wilson Score method

2. Secondary Outcome: Percentage of Participants Moderately or Strongly Preferring the Selected Treatment at Week 18 Using Question 2 of the PITPQ
Description: PITPQ Q2 was a measure of the degree of treatment preference based on the participant's opinion. The question was, "For the treatment preference you selected in Q1, what is your degree of preference?". Choices were moderate or strong.
Time Frame: Week 18
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Groups:
- Tadalafil: Participants who preferred tadalafil over sildenafil.
- Sildenafil: Participants who preferred sildenafil over tadalafil.
Arm/Group | Tadalafil | Sildenafil
Number analyzed (Participants) | 242 | 108
percentage of participants
  Strong preference | 38.0 | 34.3
  Moderate preference | 62.0 | 65.7

3. Secondary Outcome: Change in International Index of Erectile Function (IIEF) Overall Satisfaction Domain
Description: Self-reported overall satisfaction over the past 4 weeks. IIEF overall satisfaction was the sum of Q13 and Q14. Scores ranged from 1 (low/no satisfaction) to 5 (high satisfaction) for each question, with the total possible score for the 2 questions ranging from 2 to 10. Change was defined as endpoint minus baseline domain score. Change in IIEF overall satisfaction domain at Week 8 and Week 18 were averaged to produce an overall change in IIEF overall satisfaction domain score. Higher IIEF overall satisfaction domain scores were indicative of greater overall satisfaction.
Time Frame: Baseline, Week 8, and Week 18
Population: All randomized participants with baseline and at least 1 IIEF post-baseline measurement.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Tadalafil: 20 milligrams (mg) tadalafil taken orally, as needed, for 8 weeks either during Treatment Period 1 or Treatment Period 2.
- Sildenafil: 100 mg sildenafil taken orally, as needed, for 8 weeks either during Treatment Period 1 or Treatment Period 2.
Arm/Group | Tadalafil | Sildenafil
Number analyzed (Participants) | 355 | 354
units on a scale | 3.74 (1.94) | 3.71 (2.05)
Statistical Analysis 1: Comparison: Tadalafil vs Sildenafil; Test type: Superiority or Other; p = 0.793, Mixed Models Analysis — P-Value and LS mean difference were from a crossover mixed effect model that included treatment, period, sequence, and site as fixed effects, baseline value of efficacy measure as covariate, and participant within sequence as random effect; Least Squares (LS) mean difference = 0.02, 95% CI 2-sided [-0.11 to 0.15]

4. Secondary Outcome: Change in Sexual Encounter Profile (SEP) Question 2
Description: Participant-assessed diary that assessed the mean change from baseline in the percentage of "yes" responses to SEP Q2, "Were you able to insert your penis into your partner's vagina?". The SEP Q2 score was determined as the percentage of "yes" responses to SEP Q2 out of all sexual attempts recorded during the time period. Change was defined as the percentage of "yes" responses at endpoint minus the percentage of "yes" responses at baseline. Change in percentage of "yes" responses to SEP Q2 at Week 8 and Week 18 were averaged to produce an overall change in SEP Q2.
Time Frame: Baseline, Week 8, and Week 18
Population: Randomized participants with baseline and at least 1 post-baseline SEP measurement.
Measure: Mean (Standard Deviation); unit: percentage of "yes" responses
Arm/Group | Tadalafil | Sildenafil
Number analyzed (Participants) | 356 | 354
percentage of "yes" responses | 45.28 (42.03) | 44.94 (41.62)
Statistical Analysis 1: Comparison: Tadalafil vs Sildenafil; Test type: Superiority or Other; p = 0.988, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS mean difference = 0.01, 95% CI 2-sided [-1.35 to 1.37]

5. Secondary Outcome: Change in Psychosocial and Interpersonal Relationship Scale (PAIRS) Sexual Self-Confidence Domain
Description: PAIRS was a self-administered, 29-item scale that assessed the broader psychological and interpersonal outcomes associated with ED and its treatment. Each question was rated on a Likert scale that ranged from 1 (strongly disagree) to 4 (strongly agree). The sexual self-confidence domain score was the average score for Items 5, 10, 15, 23, 27, and 29. Sexual self-confidence domain scores ranged from 1 (strongly disagree) to 4 (strongly agree). Change was defined as endpoint minus baseline domain score. Change in PAIRS sexual self-confidence domain scores at Week 8 and Week 18 were averaged to produce an overall change in PAIRS sexual self-confidence domain score. Higher scores were indicative of greater sexual self-confidence.
Time Frame: Baseline, Week 8, and Week 18
Population: Randomized participants with baseline and at least 1 PAIRS post-baseline measurement.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Tadalafil: 20 mg tadalafil taken orally, as needed, for 8 weeks either during Treatment Period 1 or Treatment Period 2.
Arm/Group | Tadalafil | Sildenafil
Number analyzed (Participants) | 355 | 354
units on a scale | 0.75 (0.65) | 0.72 (0.62)
Statistical Analysis 1: Comparison: Tadalafil vs Sildenafil; Test type: Superiority or Other; p = 0.102, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS mean difference = 0.03, 95% CI 2-sided [-0.01 to 0.08]

6. Secondary Outcome: Drug Attributes Questionnaire (DRAQ) at Week 18
Description: DRAQ was a questionnaire used to record explanations for why participants preferred a drug. Participants identified their first and second reasons for drug preference from a choice of 7 reasons. Each reason for drug preference includes participants who selected that reason as their first or second reason.
Time Frame: Week 18
Population: Randomized participants who completed both treatment periods (Week 18), responded to the DRAQ, and were analyzed according to their assigned treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Tadalafil | Sildenafil
Number analyzed (Participants) | 242 | 108
percentage of participants
  Time between drug and first erection was short | 10.3 | 35.2
  Was able to get an erection long after having drug | 55.0 | 11.1
  Had erections the next morning | 24.0 | 11.1
  The firmness of erections | 36.4 | 51.9
  Was able to get an erection every time | 37.6 | 56.5
  Had few side effects | 23.6 | 25.9
  Partner preferred this treatment | 10.7 | 7.4

7. Secondary Outcome: Change in International Index of Erectile Function (IIEF) Intercourse Satisfaction Domain
Description: Self-reported intercourse satisfaction over the past 4 weeks. IIEF intercourse satisfaction was the sum of Q6, Q7, and Q8 of the IIEF. Scores ranged from 0 (low/no satisfaction) to 5 (high satisfaction) for each question, with the total possible score for the 3 questions ranging from 0 to 15. Change was defined as endpoint minus baseline domain score. Change in IIEF intercourse satisfaction domain at Week 8 and Week 18 were averaged to produce an overall change in IIEF intercourse satisfaction domain score. Higher scores were indicative of an increase in intercourse satisfaction.
Time Frame: Baseline, Week 8, and Week 18
Population: All randomized participants with baseline and at least 1 IIEF post-baseline measurement.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tadalafil | Sildenafil
Number analyzed (Participants) | 355 | 354
units on a scale | 5.88 (3.02) | 5.91 (3.03)
Statistical Analysis 1: Comparison: Tadalafil vs Sildenafil; Test type: Superiority or Other; p = 0.861, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS mean difference = -0.01, 95% CI 2-sided [-0.22 to 0.19]

8. Secondary Outcome: Change in International Index of Erectile Function (IIEF) Sexual Desire Domain
Description: Self-reported sexual desire over the past 4 weeks. IIEF sexual desire was the sum of Q11 and Q12. Scores ranged from 1 (low/almost never) to 5 (very high/almost always) for each question, with the total possible score for the 2 questions ranging from 2 to 10. Change was defined as endpoint minus baseline domain score. Change in IIEF sexual desire domain at Week 8 and Week 18 were averaged to produce an overall change in IIEF sexual desire domain score. Higher scores were indicative of increased sexual desire.
Time Frame: Baseline, Week 8, and Week 18
Population: Randomized participants with baseline and at least 1 IIEF post-baseline measurement.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tadalafil | Sildenafil
Number analyzed (Participants) | 355 | 354
units on a scale | 2.55 (2.11) | 2.60 (2.10)
Statistical Analysis 1: Comparison: Tadalafil vs Sildenafil; Test type: Superiority or Other; p = 0.495, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean Difference = -0.05, 95% CI 2-sided [-0.19 to 0.09]

9. Secondary Outcome: Change in International Index of Erectile Function (IIEF) Orgasmic Function Domain
Description: Self-reported orgasmic function over the past 4 weeks. IIEF orgasmic function was the sum of Q9 and Q10 of the IIEF. Scores ranged from 0 (no stimulation) to 5 (almost always) for each question, with the total possible score for the 2 questions ranging from 0 to 10. Change was defined as endpoint minus baseline domain score. Change in IIEF orgasmic function domain at Week 8 and Week 18 were averaged to produce an overall change in IIEF orgasmic function domain score. Higher scores were indicative of better orgasmic function.
Time Frame: Baseline, Week 8, and Week 18
Population: Randomized participants with baseline and at least 1 IIEF post-baseline measurement.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tadalafil | Sildenafil
Number analyzed (Participants) | 355 | 354
units on a scale | 3.70 (2.82) | 3.71 (2.76)
Statistical Analysis 1: Comparison: Tadalafil vs Sildenafil; Test type: Superiority or Other; p = 0.917, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS mean difference = -0.01, 95% CI 2-sided [-0.18 to 0.16]

10. Secondary Outcome: Change in Sexual Encounter Profile (SEP) Question 3
Description: Participant-assessed diary that assessed the mean change from baseline in the percentage of "yes" responses to SEP Q3, "Did your erection last long enough for you to have successful intercourse?". The SEP Q3 score was determined as the percentage of "yes" responses to SEP Q3 out of all sexual attempts recorded during the time period. Change was defined as the percentage of "yes" responses at endpoint minus percentage of "yes" responses at baseline. Change in the percentage of "yes" responses to SEP Q3 at Week 8 and Week 18 were averaged to produce an overall change in SEP Q3.
Time Frame: Baseline, Week 8, and Week 18
Population: Randomized participants with baseline and at least 1 SEP post-baseline measurement.
Measure: Mean (Standard Deviation); unit: percentage of "yes" responses
Arm/Group | Tadalafil | Sildenafil
Number analyzed (Participants) | 356 | 354
percentage of "yes" responses | 64.53 (38.37) | 63.72 (37.66)
Statistical Analysis 1: Comparison: Tadalafil vs Sildenafil; Test type: Superiority or Other; p = 0.391, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS mean difference = 1.23, 95% CI 2-sided [-1.58 to 4.04]

11. Secondary Outcome: Change in PAIRS Spontaneity Domain
Description: PAIRS was a self-administered, 29-item scale that assessed the broader psychological and interpersonal outcomes associated with ED and its treatment. Each question was rated on a Likert scale that ranged from 1 (strongly disagree) to 4 (strongly agree). The spontaneity domain score was the average score for Items 3, 12, 13, 16, 17, 19, 21, 22, and 28. Spontaneity domain scores ranged from 1 (strongly disagree) to 4 (strongly agree). Change was defined as endpoint minus baseline domain score. Change in PAIRS spontaneity domain at Week 8 and Week 18 were averaged to produce an overall change in PAIRS spontaneity domain score. Higher scores were indicative of greater spontaneity.
Time Frame: Baseline, Week 8, and Week 18
Population: Randomized participants with baseline and at least 1 PAIRS post-baseline measurement.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tadalafil | Sildenafil
Number analyzed (Participants) | 355 | 354
units on a scale | 0.33 (0.53) | 0.20 (0.42)
Statistical Analysis 1: Comparison: Tadalafil vs Sildenafil; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS mean difference = 0.13, 95% CI 2-sided [0.09 to 0.18]

12. Secondary Outcome: Change in PAIRS Time Concerns Domain
Description: PAIRS was a self-administered, 29-item scale that assessed the broader psychological and interpersonal outcomes associated with ED and its treatment. Each question was rated on a Likert scale that ranged from 1 (strongly disagree) to 4 (strongly agree). The time concerns domain score was the average score for Items 1, 2, 6, 7, 8, 20, 24, and 25. Time concern domain scores ranged from 1 (strongly disagree) to 4 (strongly agree). Change was defined as endpoint minus baseline domain score. Change in PAIRS time concerns at Week 8 and Week 18 were averaged to produce an overall change in PAIRS time concerns domain score. Higher scores were indicative of more time concerns.
Time Frame: Baseline, Week 8, and Week 18
Population: Randomized participants with baseline and at least 1 PAIRS post-baseline measurement.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tadalafil | Sildenafil
Number analyzed (Participants) | 355 | 354
units on a scale | -0.28 (0.54) | -0.14 (0.49)
Statistical Analysis 1: Comparison: Tadalafil vs Sildenafil; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS mean difference = -0.14, 95% CI 2-sided [-0.19 to -0.09]

13. Secondary Outcome: Change in International Index of Erectile Function (IIEF) Erectile Function Domain
Description: Self-reported erectile function over the past 4 weeks. IIEF erectile function was the sum of Q1 through Q5 and Q15 of the IIEF. Q1 through Q5 were scored 0 (low/no erectile function) to 5 (high erectile function) and Q15 was scored 1 (no/low confidence) to 5 (high confidence). IIEF erectile function domain scores ranged from 1 to 30. Change was defined as endpoint minus baseline domain score. Change in IIEF erectile function domain at Week 8 and Week 18 were averaged to produce an overall change in IIEF EF domain score. Higher scores were indicative of better erectile function.
Time Frame: Baseline, Week 8, and Week 18
Population: Randomized participants with baseline and at least 1 IIEF post-baseline measurement.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tadalafil | Sildenafil
Number analyzed (Participants) | 355 | 354
units on a scale | 12.03 (6.75) | 11.86 (6.68)
Statistical Analysis 1: Comparison: Tadalafil vs Sildenafil; Test type: Superiority or Other; p = 0.364, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS mean difference = 0.18, 95% CI 2-sided [-0.20 to 0.55]

ADVERSE EVENTS:
Groups:
- Tadalafil (Treatment Periods): 20 mg tadalafil taken orally, as needed, for 8 weeks either during Treatment Period 1 or Treatment Period 2.
- Sildenafil (Treatment Periods): 100 mg sildenafil taken orally, as needed, for 8 weeks either during Treatment Period 1 or Treatment Period 2.
- Tadalafil (Extension Phase): Participants who preferred tadalafil over sildenafil received 20 mg tadalafil taken orally, as needed, for an additional 8 weeks.
- Sildenafil (Extension Phase): Participants who preferred sildenafil over tadalafil received 100 mg sildenafil taken orally, as needed, for an additional 8 weeks.
Arm/Group | Tadalafil (Treatment Periods) | Sildenafil (Treatment Periods) | Tadalafil (Extension Phase) | Sildenafil (Extension Phase)
Serious Adverse Events (participants affected / at risk) | 0/363 | 0/361 | 0/231 | 0/106
Other Adverse Events (participants affected / at risk) | 30/363 | 26/361 | 7/231 | 2/106
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tadalafil (Treatment Periods) (N=363) | Sildenafil (Treatment Periods) (N=361) | Tadalafil (Extension Phase) (N=231) | Sildenafil (Extension Phase) (N=106)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Deafness (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Eye swelling (Eye disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (3) | 1 (1) | 0 (0)
Face oedema (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Feeling hot (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Thirst (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Body temperature increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 6 (7) | 3 (3) | 2 (4) | 0 (0)
Headache (Nervous system disorders) | 10 (13) | 5 (5) | 2 (4) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 3 (3) | 1 (1) | 0 (0)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 2 (2) | 6 (7) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Varicose vein (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days